CLINICAL TRIAL: NCT00157027
Title: The Use of Extracorporeal Photochemotherapy With UVADEX in Patients With HIV Who Are Refractory or Intolerant to HAART
Brief Title: RHIV A Pilot Study Refractory or Intolerant to Highly Active Antiretroviral Therapy (HAART)
Acronym: HIV-HAART
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Atlantic Health System (Other)
Collaborators: Therakos (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R03-05-012
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; HIV-1 Positive by ELISA Assay; Confirmed by Western Blot; Refractory or intolerant to HAART
MeSH Terms: conditions — HIV Infections | interventions — Photopheresis; Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Photopheresis (or extracorporeal photoimmunetherapy [ECP]) is a process developed by THERAKOS, Inc., a Johnson and Johnson Company. During the process of ECP, whole blood is drawn from the patient over several cycles, centrifuged and separated into the components of plasma, white cells (or buffy coat), and red blood cells. A portion of the white cells and the plasma are saved in a separate compartment. The remaining plasma and red blood cells are immediately returned to the patient.
  The saved buffy coat (white blood cells) and plasma are inoculated with the photosensitizing agent UVADEX. Photoactivation begins when the suspension is exposed to a prescribed amount of ultraviolet-A light. After photoactivation is complete, the treated suspension is returned to the patient.
  Interventions: Procedure: Extracorporeal photochemotherapy with UVADEX

INTERVENTIONS:
Procedure: Extracorporeal photochemotherapy with UVADEX — Photopheresis (or extracorporeal photoimmunetherapy [ECP]) is a process developed by THERAKOS, Inc., a Johnson and Johnson Company. During the process of ECP, whole blood is drawn from the patient over several cycles, centrifuged and separated into the components of plasma, white cells (or buffy coat), and red blood cells. A portion of the white cells and the plasma are saved in a separate compartment. The remaining plasma and red blood cells are immediately returned to the patient.
  The saved buffy coat (white blood cells) and plasma are inoculated with the photosensitizing agent UVADEX. Photoactivation begins when the suspension is exposed to a prescribed amount of ultraviolet-A light. After photoactivation is complete, the treated suspension is returned to the patient.

SUMMARY:
The objectives of this clinical trial are to:

* Assess the safety of using extracorporeal photoimmune therapy with the photosensitizing agent Uvadex in the treatment of HIV-1 infection;
* Evaluate the effects of this therapy on HIV-1 viral load by polymerase chain reaction (PCR) analysis;
* Evaluate the effects of this therapy on CD4+, CD8+ cells and CD4/CD8 ratio;
* Evaluate the effects of this therapy on the patient's immune system, by skin reactivity to a standard anergy panel.

DETAILED DESCRIPTION:
Rationale for the Use of ECP with UVADEX in Patients with HIV-1 Infection

Studies have demonstrated that psoralen and ultraviolet A light inactivate HIV virus in vitro. Edelson, et al, showed that extracorporeal photochemotherapy (ECP) with psoralen primarily targets the CD4+ cell, the population predominately affected by HIV-1 infection. It is postulated that the re-infusion of the ECP treated cell fraction, free virus, cell-associated virus along with whole cells, cell fragments, and soluble antigens, may serve to engender a specific HIV immune response.

A twenty-patient study using ECP with psoralen was conducted by Bisaccia, et al. In this study, patients were HIV positive by enzyme linked immunosorbent assay and these positive results were confirmed by Western blot test. Patients were staged as Walter Reed class WR3 to WR5. Extracorporeal photoimmune therapy was administered on two consecutive days on a monthly basis for 6-29 months. This study reported that CD4 counts declined more slowly than historical controls. Walter Reed classification improved in 55% (11/20), was stable in 35% (7/20) and declined in 10% (2/20) of the patients treated in this study.

One measure in the "in vivo" evaluation of T-cell function is provided by skin reactivity to recall antigens (DTH). A lack of this response has been associated with progression of HIV disease. In the Bisaccia study, skin reactivity to recall antigens (DTH) improved in 55% (11/20) patients, were stable in 35% (7/20), progressed to anergy in 5% (1/20). One patient was initially anergic and remained anergic post-treatment. Following treatment with ECP, 60% (9/15), displayed normal skin test responses, whereas the baseline examinations had been normal in only 5% (1/19). In addition, 21% (4/19) of patients showed a partial skin test response. Only 10% (2/20) of patients developed a new opportunistic infection. This included the patient initially anergic and who remained anergic and the patient who progressed to anergy post-ECP treatment.

DESCRIPTION OF THE UVAR® XTSÔ PHOTOPHERESIS SYSTEM

Photopheresis (or extracorporeal photoimmune therapy [ECP]) is a process developed by THERAKOS, Inc., a Johnson and Johnson Company. During the process of ECP, whole blood is drawn from the patient over several cycles, centrifuged and separated into the components of plasma, white cells (or buffy coat), and red blood cells. A portion of the white cells and the plasma are saved in a separate compartment. The remaining plasma and red blood cells are immediately returned to the patient.

The saved buffy coat (white blood cells) and plasma are inoculated with the photosensitizing agent UVADEX. Photoactivation begins when the suspension is exposed to a prescribed amount of ultraviolet-A light. After photoactivation is complete, the treated suspension is returned to the patient.

Photopheresis performed using the UVAR XTS is a continuous process. During the entire therapy, the patient remains connected to the photopheresis instrument. The duration of time between completion of the buffy coat collection and reinfusion of the light-activated buffy coat is approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive by ELISA assay and confirmed by Western blot
* Patients must be refractory or intolerant to HAART. Refractory HIV patients are defined as those patients meeting the following criteria:

  * Resistance to all major groups of active agents (non-nucleotide reverse transcriptase inhibitors [NNRTIs], nucleotide reverse transcriptase inhibitors [NRTIs], and protease inhibitors [PIs]);
  * Not achieving < 400 copies/mL by 24 weeks or < 50 copies/mL by 48 weeks of therapy; or
  * Documentation of resistance mutations by genotype testing; or
  * Failure to increase CD4+ cells > 25 cells/mm3 above baseline after one year of therapy.
* HIV RNA >= 3,000 copies/mL by PCR analysis
* CD4 count > 75 cells/mm3
* No new antiretroviral agents may be added during the pre-study evaluation, treatment, or follow-up periods.
* Life expectancy > 6 months
* Able to give informed consent and comply with all study visits, procedures, and the ECP treatment schedule
* Ages between 18 and 70
* Females of childbearing potential may not be lactating and must be human chorionic gonadotropin (HCG) negative at study entry and agree to use acceptable methods of birth control (hormonal, intrauterine device, and spermicide and barrier) throughout the study period.
* Minimum body weight of 88 lbs (40kg)
* May not have current photosensitive diseases such as systemic lupus erythematosus (SLE) or porphyria
* Adequate hematological function with an absolute neutrophil count of >= 500/mm and a platelet count of >= 50,000/mm.

Exclusion Criteria:

* Established history of heparin or psoralen allergy
* Patients with aphakia because of significantly increased risk of retinal damage due to absence of lenses. Patients with lens implants are acceptable for inclusion.
* Current participation (within 30 days) in a clinical trial examining the safety and/or efficacy of anti-retroviral agent(s)
* Patients with any other major illness (e.g. malignancy, renal failure, severe cardiac disease, severe neurologic disease) that either might preclude completion of the study or bias efficacy assessments.
* Patients who cannot or may not tolerate the extracorporeal volume required during the procedure, for reasons such as severe cardiovascular disease, i.e. history of congestive heart failure or severe anemia (hemoglobin < 90 g/L)
* Patients with a photosensitive disease, such as porphyria or systemic lupus erythematosus. Special care must be taken in the treatment of patients who require medications (either topically or systemically) during the course of the study with photosensitizing potential, such as phenothiazine, tetracyclines, sulfonamides, some non-steroidal anti-inflammatory drugs (NSAIDs) or chlorothiazide. Patients who must take photosensitizing drugs during the study will not receive them within 24 hours of each scheduled treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-12; Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
evaluate the effects of this therapy on HIV-1 viral load by PCR analysis | 9 months
evaluate the effects of this therapy on CD4+, CD8+ cells and CD4/CD8 ratio | 9 months
evaluate the effects of this therapy on the patient's immune system, by skin reactivity to a standard anergy panel | 9 months
The objectives of this clinical trial are to: assess the safety of using extracorporeal photoimmune therapy with the photosensitizing agent UVADEX in the treatment of HIV-1 infection. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Emil Bisaccia, MD, Principal Investigator — Morristown Memorial Hospital-Atlantic Health System